CLINICAL TRIAL: NCT02927873
Title: A Phase 1/2, Randomized, Observer-blind, Controlled, Multi-center, Dose-escalation Study to Evaluate Safety, Reactogenicity and Immunogenicity of GSK Biologicals' Respiratory Syncytial Virus (RSV) Investigational Vaccine Based on the RSV Viral Proteins F, N and M2-1 Encoded by Chimpanzee-derived Adenovector (ChAd155-RSV) (GSK3389245A), When Administered Intramuscularly According to a 0, 1-month Schedule to RSV-seropositive Infants Aged 12 to 23 Months
Brief Title: A Study to Evaluate Safety, Reactogenicity and Immunogenicity of GSK Biologicals' RSV Investigational Vaccine Based on Viral Proteins Encoded by Chimpanzee-derived Adenovector (ChAd155-RSV) (GSK3389245A) in RSV-seropositive Infants
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 204838; 2016-000117-76 (EudraCT Number)
Record Dates: First submitted 2016-10-06; First posted 2016-10-07 (Estimated); Results first posted 2021-10-28 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-09

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Safety; Respiratory syncytial virus (RSV); Immunogenicity; Reactogenicity; Infants; Vaccine
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Observer blind
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- RSV LD Group (Experimental): RSV-seropositive infants, aged 12 to 23 months at the time of first vaccination, received 2 doses (0.5 mL each) of the RSV low dose (LD) vaccine, administered intramuscularly, one each at Day 1 and Day 31.
  Interventions: Biological: RSV (GSK3389245A) low dose formulation vaccine
- RSV MD Group (Experimental): RSV-seropositive infants, aged 12 to 23 months at the time of first vaccination, received 2 doses (0.15 mL each) of the RSV middle dose (MD) vaccine, administered intramuscularly, one each at Day 1 and Day 31.
  Interventions: Biological: RSV (GSK3389245A) middle dose formulation vaccine
- RSV HD Group (Experimental): RSV-seropositive infants, aged 12 to 23 months at the time of first vaccination, received 2 doses (0.5 mL each) of the RSV high dose (HD) vaccine, administered intramuscularly, one each at Day 1 and Day 31.
  Interventions: Biological: RSV (GSK3389245A) high dose formulation vaccine
- Placebo LD group (Placebo Comparator): RSV-seropositive infants, aged 12 to 23 months at the time of first vaccination, received 2 doses (0.5 mL each) of placebo, administered intramuscularly, one each at Day 1 and Day 31.
  Interventions: Drug: Placebo
- Placebo MD group (Placebo Comparator): RSV-seropositive infants, aged 12 to 23 months at the time of first vaccination, received 2 doses (0.15 mL each) of placebo, administered intramuscularly, one each at Day 1 and Day 31.
  Interventions: Drug: Placebo
- Placebo HD group (Placebo Comparator): RSV-seropositive infants, aged 12 to 23 months at the time of first vaccination, received 2 doses (0.5 mL each) of placebo, administered intramuscularly, one each at Day 1 and Day 31.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: RSV (GSK3389245A) low dose formulation vaccine — 2 doses of 0.5 ml each of RSV (GSK3389245A) low dose formulation vaccine administered intramuscularly in the left anterolateral thigh or deltoid, at Day 1 and Day 31.
  Arms: RSV LD Group
Biological: RSV (GSK3389245A) middle dose formulation vaccine — 2 doses of 0.15 ml each of RSV (GSK3389245A) middle dose formulation vaccine administered intramuscularly in the left anterolateral thigh or deltoid, at Day 1 and Day 31.
  Arms: RSV MD Group
Biological: RSV (GSK3389245A) high dose formulation vaccine — 2 doses of 0.5 ml each of RSV (GSK3389245A) high dose formulation vaccine administered intramuscularly in the left anterolateral thigh or deltoid, at Day 1 and Day 31.
  Arms: RSV HD Group
Drug: Placebo — 2 doses (0.5 mL each for Placebo LD and Placebo HD groups and 0.15 mL each for Placebo MD group) of Placebo administered intramuscularly in the left anterolateral thigh or deltoid, at Day 1 and Day 31.
  Arms: Placebo HD group; Placebo LD group; Placebo MD group

SUMMARY:
The purpose of this study is to evaluate the safety, reactogenicity and immunogenicity of the respiratory syncytial virus (RSV) candidate vaccine when first administered via intramuscular (IM) injection according to a 0, 1-month schedule to RSV-seropositive infants aged 12 to 23 months.

DETAILED DESCRIPTION:
The RSV PED-002 study, designed to evaluate the safety, reactogenicity and immunogenicity of the RSV candidate vaccine when administered in 3 sequential doses to seropositive infants aged 12 to 23 months, will be conducted in an observer-blind manner in Epoch 1 and single-blinded in Epoch 2.

ELIGIBILITY:
Inclusion Criteria:

* Subjects' parent(s)/ Legally acceptable representative (LAR[s]) who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written informed consent obtained from the parent(s)/LAR(s) of the subject prior to performance of any study specific procedure.
* A male or female between, and including, 12 and 23 months at the time of the first vaccination.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Seropositive for RSV as determined by IBL International kit.
* Born full-term (i.e. after a gestation period of 37 to less than 42 completed weeks) with a minimum birth weight of 2.5 kg. (Required for Spain)
* Subjects' parent(s)/LAR(s) need to have access to a consistent mean of telephone contact or computer.

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product other than the study vaccine during the period starting 30 days before the first dose of study vaccine (Day -29 to Day 0), or planned use during the study period.
* Any medical condition that in the judgment of the investigator would make IM injection unsafe.
* Chronic administration of immunosuppressants or other immune-modifying drugs during the period starting six months prior to the first vaccine. For corticosteroids, this will mean prednisone, or equivalent. Inhaled and topical steroids are allowed.
* Administration of long-acting immune-modifying drugs or planned administration at any time during the study period.
* Administration of immunoglobulins and/or any blood products during the period starting three months before the first dose of study vaccine or planned administration during the study period.
* Planned administration/administration of a vaccine not foreseen by the study protocol in the period starting 30 days before the first dose and ending 30 days after the last dose of vaccine administration, with the exception of scheduled routine pediatric vaccines which may be administered ≥ 14 days before a dose or ≥ 7 days after a dose.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Serious chronic illness.
* Major congenital defects.
* History of any neurological disorders or seizures.
* History of or current autoimmune disease.
* History of recurrent wheezing.
* History of chronic cough.
* Previous hospitalization for respiratory illnesses.
* History of thrombocytopenia.
* History of anemia.
* Previous, current or planned administration of Synagis.
* Neurological complications following any prior vaccination.
* Born to a mother known or suspected to be HIV-positive.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Family history of congenital or hereditary immunodeficiency.
* Previous vaccination with a recombinant simian or human adenoviral vaccine.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* Hypersensitivity to latex.
* Current severe eczema.
* Acute disease and/or fever at the time of enrolment.

  * Fever is defined as temperature ≥ 37.5°C/99.5°F for oral, axillary or tympanic route, or ≥ 38.0°C/100.4°F for rectal route. The preferred route for recording temperature in this study will be axillary.
  * Clinically significant upper respiratory tract infection
  * Subjects with a minor illness without fever may, be enrolled at the discretion of the investigator.
* Any clinically significant Grade 1 or any ≥ Grade 2 hematological or biochemical laboratory abnormality detected at the last screening blood sampling.
* Any other conditions that the investigator judges may interfere with study procedures or findings.
* Any conditions that could constitute a risk for the subjects while participating to this study.
* Weight below the fifth percentile of the local weight-for-age curve.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product.
* Planned move to a location that will prohibit participating in the trial until study end.

Ages: 12 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 107 (Actual)
Dates: Start 2017-01-11 (Actual); Primary Completion 2019-02-19 (Actual); Study Completion 2020-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (21):
- United States (6):
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, Frederick, Maryland
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Sioux Falls, South Dakota
- GSK Investigational Site, Halifax, Nova Scotia, Canada
- Italy (2):
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Perugia, Umbria
- GSK Investigational Site, México, Mexico
- Panama (2):
  - GSK Investigational Site, David, Chiriquí Province
  - GSK Investigational Site, Panama City
- GSK Investigational Site, Dębica, Poland
- Spain (5):
  - GSK Investigational Site, Burgos
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Majadahonda (Madrid)
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Valencia
- Taiwan (3):
  - GSK Investigational Site, Hsinchu
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Diez-Domingo J, Saez-Llorens X, Rodriguez-Weber MA, Epalza C, Chatterjee A, Chiu CH, Lin CY, Berry AA, Martinon-Torres F, Baquero-Artigao F, Langley JM, Ramos Amador JT, Domachowske JB, Huang LM, Chiu NC, Esposito S, Moris P, Lien-Anh Nguyen T, Nikic V, Woo W, Zhou Y, Dieussaert I, Leach A, Gonzalez Lopez A, Vanhoutte N. Safety and Immunogenicity of a ChAd155-Vectored Respiratory Syncytial Virus (RSV) Vaccine in Healthy RSV-Seropositive Children 12-23 Months of Age. J Infect Dis. 2023 May 29;227(11):1293-1302. doi: 10.1093/infdis/jiac481. PMID 36484484

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 32 centers in 8 countries (Canada, Italy, Mexico, Panama, Poland, Spain, Taiwan and United States).
Pre-assignment Details: Out of 107 participants enrolled in the study, 21 participants were not assigned to any study group and 4 participants did not receive any study treatment.
  82 subjects were vaccinated and included in the Exposed Set.
Period: Overall Study
Arm/Group | RSV LD Group | RSV MD Group | RSV HD Group | Placebo LD Group | Placebo MD Group | Placebo HD Group
Started | 11 | 14 | 18 | 11 | 11 | 17
Completed | 9 | 11 | 18 | 11 | 11 | 16
Not Completed | 2 | 3 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0
Not completed — CONSENT WITHDRAWAL NOT DUE TO ADV. EVENT | 0 | 1 | 0 | 0 | 0 | 0
Not completed — MIGRATED / MOVED FROM THE STUDY AREA | 0 | 0 | 0 | 0 | 0 | 1
Not completed — PARENTS NOT ABLE TO COME TO SITE | 0 | 1 | 0 | 0 | 0 | 0
Not completed — SUBJECT WITHDRAWN AT AN INTERIM TIMEPOINT, BUT ACCEPTED CALLS FOR SAFETY SURVEILLANCE | 1 | 0 | 0 | 0 | 0 | 0
Not completed — PARENTS REFUSED SAFETY FOLLOW-UP | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RSV LD Group | RSV MD Group | RSV HD Group | Placebo LD Group | Placebo MD Group | Placebo HD Group | Total
Number analyzed (Participants) | 11 | 14 | 18 | 11 | 11 | 17 | 82
Age, Continuous [Mean (Standard Deviation); unit: MONTHS] | 15.4 (1.6) | 15.6 (3.3) | 16.3 (4.0) | 15.0 (1.9) | 16.2 (2.7) | 17.4 (3.8) | 16.1 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 10 | 5 | 3 | 12 | 41
  Male | 7 | 7 | 8 | 6 | 8 | 5 | 41
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  AFRICAN HERITAGE / AFRICAN AMERICAN | 0 | 0 | 0 | 0 | 1 | 0 | 1
  ASIAN - EAST ASIAN HERITAGE | 0 | 0 | 3 | 0 | 1 | 3 | 7
  ASIAN - SOUTH EAST ASIAN HERITAGE | 0 | 0 | 1 | 0 | 1 | 0 | 2
  NATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER | 0 | 1 | 0 | 0 | 0 | 0 | 1
  OTHER, NOT SPECIFIED | 0 | 7 | 12 | 2 | 4 | 9 | 34
  WHITE - CAUCASIAN / EUROPEAN HERITAGE | 11 | 6 | 2 | 9 | 4 | 5 | 37

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Any Solicited Local Adverse Events (AEs)
Description: Assessed solicited local symptoms are pain, redness and swelling at injection site. Any = occurrence of the symptom regardless of intensity grade. Any redness and swelling symptom = symptom reported with a surface diameter greater than 0 millimeters.
Time Frame: During a 7-day follow-up period after each vaccination (vaccine/placebo administered at Day 1 and Day 31)
Population: This analysis was performed on the Exposed Set, which included all subjects with at least one study vaccine administration documented and with the diary card completed after each vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV LD Group | RSV MD Group | RSV HD Group | Placebo LD Group | Placebo MD Group | Placebo HD Group
Number analyzed (Participants) | 11 | 13 | 18 | 11 | 11 | 17
Participants
  DOSE 1, Any Pain | 1 | 2 | 0 | 2 | 0 | 2
  DOSE 1, Any Redness | 2 | 1 | 3 | 3 | 0 | 3
  DOSE 1, Any Swelling | 0 | 0 | 1 | 1 | 1 | 2
  DOSE 2, Any Pain: number analyzed (Participants) | 10 | 12 | 17 | 11 | 11 | 17
  DOSE 2, Any Pain | 2 | 2 | 2 | 1 | 0 | 3
  DOSE 2, Any Redness: number analyzed (Participants) | 10 | 12 | 17 | 11 | 11 | 17
  DOSE 2, Any Redness | 2 | 1 | 2 | 3 | 0 | 2
  DOSE 2, Any Swelling: number analyzed (Participants) | 10 | 12 | 17 | 11 | 11 | 17
  DOSE 2, Any Swelling | 0 | 0 | 0 | 1 | 0 | 2

2. Primary Outcome: Number of Subjects With Any Solicited General AEs
Description: Assessed solicited general symptoms are drowsiness, fever [defined as temperature equal to or above (≥) 37.5 degrees Celsius (°C)/99.5 degrees Fahrenheit (°F) for oral, axillary or tympanic route, or ≥ 38.0°C/100.4°F for rectal route, the preferred route for recording temperature in this study being axillary], irritability/fussiness and loss of appetite. Any = occurrence of the symptom regardless of intensity grade or relation to study vaccination.
Time Frame: During a 7-day follow-up period after each vaccination (vaccine/placebo administered at Day 1 and Day 31)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | RSV LD Group | RSV MD Group | RSV HD Group | Placebo LD Group | Placebo MD Group | Placebo HD Group
Number analyzed (Participants) | 11 | 13 | 18 | 11 | 11 | 17
Participants
  DOSE 1, Any Drowsiness | 4 | 2 | 4 | 5 | 3 | 4
  DOSE 1, Any Irritability / Fussiness | 3 | 3 | 4 | 4 | 2 | 2
  DOSE 1, Any Loss Of Appetite | 3 | 3 | 4 | 2 | 2 | 3
  DOSE 1, Any Fever | 3 | 3 | 10 | 3 | 2 | 0
  DOSE 2, Any Drowsiness: number analyzed (Participants) | 10 | 12 | 17 | 11 | 11 | 17
  DOSE 2, Any Drowsiness | 2 | 1 | 5 | 3 | 2 | 5
  DOSE 2, Any Irritability / Fussiness: number analyzed (Participants) | 10 | 12 | 17 | 11 | 11 | 17
  DOSE 2, Any Irritability / Fussiness | 3 | 1 | 5 | 3 | 1 | 6
  DOSE 2, Any Loss Of Appetite: number analyzed (Participants) | 10 | 12 | 17 | 11 | 11 | 17
  DOSE 2, Any Loss Of Appetite | 3 | 0 | 6 | 3 | 2 | 5
  DOSE 2, Any Fever: number analyzed (Participants) | 10 | 12 | 17 | 11 | 11 | 17
  DOSE 2, Any Fever | 2 | 2 | 5 | 1 | 2 | 1

3. Primary Outcome: Number of Subjects With Any Unsolicited AEs
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Unsolicited AEs are reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any is defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to study vaccination.
Time Frame: During a 30-day follow-up period after each vaccination (vaccine/placebo administered at Day 1 and Day 31)
Population: This analysis was performed on the Exposed Set, which included all subjects with at least one study vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV LD Group | RSV MD Group | RSV HD Group | Placebo LD Group | Placebo MD Group | Placebo HD Group
Number analyzed (Participants) | 11 | 14 | 18 | 11 | 11 | 17
Participants | 9 | 9 | 13 | 7 | 10 | 13

4. Primary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs) From Day 1 up to Day 61
Description: Assessed SAEs include any untoward medical occurrences that resulted in death, were life-threatening, required hospitalization or prolongation of hospitalization or resulted in disability/incapacity. Any = occurrence of SAE regardless of intensity grade or relation to study vaccination.
Time Frame: From Day 1 up to Day 61
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | RSV LD Group | RSV MD Group | RSV HD Group | Placebo LD Group | Placebo MD Group | Placebo HD Group
Number analyzed (Participants) | 11 | 14 | 18 | 11 | 11 | 17
Participants | 0 | 0 | 1 | 1 | 0 | 2

5. Primary Outcome: Number of Subjects With Episode of Spontaneous or Excessive Bleeding (AE of Specific Interest)
Description: Any episode of spontaneous or excessive bleeding if occurring after vaccination was to be fully investigated with a full range of hematological tests to identify the underlying cause and reported as an AE of specific interest.
Time Frame: During a 30-day follow-up period after each vaccination (vaccine/placebo administered at Day 1 and Day 31)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | RSV LD Group | RSV MD Group | RSV HD Group | Placebo LD Group | Placebo MD Group | Placebo HD Group
Number analyzed (Participants) | 11 | 14 | 18 | 11 | 11 | 17
Participants | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Subjects With Hematological Laboratory Results Change With Respect to Normal Laboratory Ranges and Versus Baseline, at Day 2
Description: Assessed hematological laboratory parameters include hemoglobin level [HgL] white blood cells [WBC] and platelet count [PLC]. Hematological abnormalities refer to range indicator at timing, categorized as Below, Within or Above normal ranges, and compared to baseline range indicator of the same parameter, at Screening (Day-29 to Day 1) i.e. Unknown, Below, Within or Above. [e.g. HgL, Below, Below = HgL below normal ranges at baseline versus below normal ranges at Day 2].
Time Frame: At Day 2
Population: This analysis was performed on the Exposed Set, which included all subjects with at least one study vaccine administration documented and with available results for the specified parameter and time point.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV LD Group | RSV MD Group | RSV HD Group | Placebo LD Group | Placebo MD Group | Placebo HD Group
Number analyzed (Participants) | 11 | 14 | 15 | 11 | 11 | 16
Participants
  HgL, Below, Below: number analyzed (Participants) | 3 | 2 | 1 | 1 | 0 | 0
  HgL, Below, Below | 3 | 2 | 1 | 1 | 0 | 0
  HgL, Within, Unknown: number analyzed (Participants) | 8 | 12 | 15 | 10 | 11 | 16
  HgL, Within, Unknown | 0 | 1 | 0 | 0 | 0 | 0
  HgL, Within, Below: number analyzed (Participants) | 8 | 12 | 15 | 10 | 11 | 16
  HgL, Within, Below | 0 | 2 | 0 | 0 | 2 | 2
  HgL, Within, Within: number analyzed (Participants) | 8 | 12 | 15 | 10 | 11 | 16
  HgL, Within, Within | 8 | 9 | 15 | 10 | 9 | 13
  HgL, Within, Above: number analyzed (Participants) | 8 | 12 | 15 | 10 | 11 | 16
  HgL, Within, Above | 0 | 0 | 0 | 0 | 0 | 1
  HgL, Above, Within: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 1
  HgL, Above, Within | 0 | 0 | 0 | 0 | 0 | 1
  HgL, Above, Above: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 1
  HgL, Above, Above | 0 | 0 | 1 | 0 | 0 | 0
  WBC, Below, Below: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 1
  WBC, Below, Below | 0 | 0 | 1 | 0 | 0 | 0
  WBC, Below, Within: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 1
  WBC, Below, Within | 0 | 0 | 0 | 0 | 0 | 1
  WBC, Within, Unknown: number analyzed (Participants) | 11 | 14 | 14 | 11 | 7 | 16
  WBC, Within, Unknown | 0 | 1 | 0 | 0 | 0 | 0
  WBC, Within, Below: number analyzed (Participants) | 11 | 14 | 14 | 11 | 7 | 16
  WBC, Within, Below | 0 | 2 | 1 | 0 | 0 | 2
  WBC, Within, Within: number analyzed (Participants) | 11 | 14 | 14 | 11 | 7 | 16
  WBC, Within, Within | 11 | 11 | 13 | 11 | 6 | 13
  WBC, Within, Above: number analyzed (Participants) | 11 | 14 | 14 | 11 | 7 | 16
  WBC, Within, Above | 0 | 0 | 0 | 0 | 1 | 1
  WBC, Above, Within: number analyzed (Participants) | 0 | 0 | 2 | 0 | 4 | 0
  WBC, Above, Within | 0 | 0 | 1 | 0 | 2 | 0
  WBC, Above, Above: number analyzed (Participants) | 0 | 0 | 2 | 0 | 4 | 0
  WBC, Above, Above | 0 | 0 | 1 | 0 | 2 | 0
  PLC, Within, Unknown: number analyzed (Participants) | 10 | 12 | 15 | 9 | 6 | 15
  PLC, Within, Unknown | 0 | 1 | 0 | 0 | 0 | 0
  PLC, Within, Below: number analyzed (Participants) | 10 | 12 | 15 | 9 | 6 | 15
  PLC, Within, Below | 0 | 0 | 1 | 0 | 0 | 0
  PLC, Within, Within: number analyzed (Participants) | 10 | 12 | 15 | 9 | 6 | 15
  PLC, Within, Within | 10 | 10 | 12 | 9 | 4 | 12
  PLC, Within, Above: number analyzed (Participants) | 10 | 12 | 15 | 9 | 6 | 15
  PLC, Within, Above | 0 | 1 | 2 | 0 | 2 | 3
  PLC, Above, Within: number analyzed (Participants) | 1 | 1 | 2 | 2 | 5 | 2
  PLC, Above, Within | 1 | 1 | 2 | 1 | 2 | 0
  PLC, Above, Above: number analyzed (Participants) | 1 | 1 | 2 | 2 | 5 | 2
  PLC, Above, Above | 0 | 0 | 0 | 1 | 3 | 2

7. Primary Outcome: Number of Subjects With Hematological Laboratory Results Change With Respect to Normal Laboratory Ranges and Versus Baseline, at Day 8
Description: Assessed hematological laboratory parameters include hemoglobin level [HgL] white blood cells [WBC] and platelet count [PLC]. Hematological abnormalities refer to range indicator at timing, categorized as Below, Within or Above normal ranges, and compared to baseline range indicator of the same parameter, at Screening (Day-29 to Day 1) i.e. Below, Within or Above. [e.g. HgL, Below, Below = HgL below normal ranges at baseline versus below normal ranges at Day 8].
Time Frame: At Day 8
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | RSV LD Group | RSV MD Group | RSV HD Group | Placebo LD Group | Placebo MD Group | Placebo HD Group
Number analyzed (Participants) | 9 | 3 | 2 | 8 | 5 | 3
Participants
  HgL, Below, Below: number analyzed (Participants) | 2 | 1 | 0 | 1 | 0 | 0
  HgL, Below, Below | 2 | 1 | 0 | 1 | 0 | 0
  HgL, Within, Within: number analyzed (Participants) | 7 | 2 | 2 | 7 | 5 | 2
  HgL, Within, Within | 7 | 2 | 2 | 7 | 5 | 2
  HgL, Above, Above: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  HgL, Above, Above | 0 | 0 | 0 | 0 | 0 | 1
  WBC, Within, Within: number analyzed (Participants) | 9 | 3 | 2 | 8 | 2 | 3
  WBC, Within, Within | 8 | 2 | 2 | 8 | 2 | 3
  WBC, Within, Above: number analyzed (Participants) | 9 | 3 | 2 | 8 | 2 | 3
  WBC, Within, Above | 1 | 1 | 0 | 0 | 0 | 0
  WBC, Above, Within: number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 0
  WBC, Above, Within | 0 | 0 | 0 | 0 | 3 | 0
  PLC, Within, Within: number analyzed (Participants) | 8 | 3 | 2 | 8 | 3 | 3
  PLC, Within, Within | 7 | 3 | 1 | 8 | 0 | 3
  PLC, Within, Above: number analyzed (Participants) | 8 | 3 | 2 | 8 | 3 | 3
  PLC, Within, Above | 1 | 0 | 1 | 0 | 3 | 0
  PLC, Above, Within: number analyzed (Participants) | 1 | 0 | 0 | 0 | 2 | 0
  PLC, Above, Within | 1 | 0 | 0 | 0 | 1 | 0
  PLC, Above, Above: number analyzed (Participants) | 1 | 0 | 0 | 0 | 2 | 0
  PLC, Above, Above | 0 | 0 | 0 | 0 | 1 | 0

8. Primary Outcome: Number of Subjects With Hematological Laboratory Results Change With Respect to Normal Laboratory Ranges and Versus Baseline, at Day 31
Description: Assessed hematological laboratory parameters include hemoglobin level [HgL] white blood cells [WBC] and platelet count [PLC]. Hematological abnormalities refer to range indicator at timing, categorized as Below, Within or Above normal ranges, and compared to baseline range indicator of the same parameter, at Screening (Day-29 to Day 1) i.e. Unknown, Below, Within or Above. [e.g. HgL, Below, Below = HgL below normal ranges at baseline versus below normal ranges at Day 31].
Time Frame: At Day 31
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | RSV LD Group | RSV MD Group | RSV HD Group | Placebo LD Group | Placebo MD Group | Placebo HD Group
Number analyzed (Participants) | 10 | 12 | 16 | 10 | 9 | 16
Participants
  HgL, Below, Below: number analyzed (Participants) | 3 | 2 | 1 | 1 | 0 | 0
  HgL, Below, Below | 3 | 1 | 1 | 1 | 0 | 0
  HgL, Below, Within: number analyzed (Participants) | 3 | 2 | 1 | 1 | 0 | 0
  HgL, Below, Within | 0 | 1 | 0 | 0 | 0 | 0
  HgL, Within, Unknown: number analyzed (Participants) | 7 | 10 | 16 | 9 | 9 | 16
  HgL, Within, Unknown | 0 | 1 | 0 | 0 | 0 | 0
  HgL, Within, Below: number analyzed (Participants) | 7 | 10 | 16 | 9 | 9 | 16
  HgL, Within, Below | 0 | 0 | 0 | 0 | 1 | 2
  HgL, Within, Within: number analyzed (Participants) | 7 | 10 | 16 | 9 | 9 | 16
  HgL, Within, Within | 7 | 9 | 15 | 9 | 8 | 14
  HgL, Within, Above: number analyzed (Participants) | 7 | 10 | 16 | 9 | 9 | 16
  HgL, Within, Above | 0 | 0 | 1 | 0 | 0 | 0
  HgL, Above, Within: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 1
  HgL, Above, Within | 0 | 0 | 1 | 0 | 0 | 1
  WBC, Below, Within: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 1
  WBC, Below, Within | 0 | 0 | 1 | 0 | 0 | 1
  WBC, Within, Unknown: number analyzed (Participants) | 10 | 12 | 15 | 10 | 5 | 16
  WBC, Within, Unknown | 0 | 1 | 0 | 0 | 0 | 0
  WBC, Within, Below: number analyzed (Participants) | 10 | 12 | 15 | 10 | 5 | 16
  WBC, Within, Below | 0 | 0 | 0 | 0 | 0 | 1
  WBC, Within, Within: number analyzed (Participants) | 10 | 12 | 15 | 10 | 5 | 16
  WBC, Within, Within | 10 | 9 | 13 | 10 | 4 | 15
  WBC, Within, Above: number analyzed (Participants) | 10 | 12 | 15 | 10 | 5 | 16
  WBC, Within, Above | 0 | 2 | 2 | 0 | 1 | 0
  WBC, Above, Within: number analyzed (Participants) | 0 | 0 | 2 | 0 | 4 | 0
  WBC, Above, Within | 0 | 0 | 1 | 0 | 3 | 0
  WBC, Above, Above: number analyzed (Participants) | 0 | 0 | 2 | 0 | 4 | 0
  WBC, Above, Above | 0 | 0 | 1 | 0 | 1 | 0
  PLC, Within, Unknown: number analyzed (Participants) | 10 | 11 | 16 | 8 | 5 | 15
  PLC, Within, Unknown | 0 | 1 | 0 | 0 | 0 | 0
  PLC, Within, Within: number analyzed (Participants) | 10 | 11 | 16 | 8 | 5 | 15
  PLC, Within, Within | 9 | 8 | 15 | 8 | 4 | 13
  PLC, Within, Above: number analyzed (Participants) | 10 | 11 | 16 | 8 | 5 | 15
  PLC, Within, Above | 1 | 2 | 1 | 0 | 1 | 2
  PLC, Above, Within: number analyzed (Participants) | 0 | 1 | 2 | 2 | 4 | 2
  PLC, Above, Within | 0 | 1 | 2 | 2 | 2 | 1
  PLC, Above, Above: number analyzed (Participants) | 0 | 1 | 2 | 2 | 4 | 2
  PLC, Above, Above | 0 | 0 | 0 | 0 | 2 | 1

9. Primary Outcome: Number of Subjects With Hematological Laboratory Results Change With Respect to Normal Laboratory Ranges and Versus Baseline, at Day 32
Description: Assessed hematological laboratory parameters include hemoglobin level [HgL] white blood cells [WBC] and platelet count [PLC]. Hematological abnormalities refer to range indicator at timing, categorized as Below, Within or Above normal ranges, and compared to baseline range indicator of the same parameter, at Screening (Day-29 to Day 1) i.e. Unknown, Below, Within or Above. [e.g. HgL, Below, Below = HgL below normal ranges at baseline versus below normal ranges at Day 32].
Time Frame: At Day 32
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | RSV LD Group | RSV MD Group | RSV HD Group | Placebo LD Group | Placebo MD Group | Placebo HD Group
Number analyzed (Participants) | 10 | 10 | 15 | 11 | 10 | 16
Participants
  HgL, Below, Below: number analyzed (Participants) | 3 | 2 | 1 | 1 | 0 | 0
  HgL, Below, Below | 2 | 2 | 1 | 1 | 0 | 0
  HgL, Below, Within: number analyzed (Participants) | 3 | 2 | 1 | 1 | 0 | 0
  HgL, Below, Within | 1 | 0 | 0 | 0 | 0 | 0
  HgL, Within, Unknown: number analyzed (Participants) | 7 | 8 | 15 | 10 | 10 | 16
  HgL, Within, Unknown | 0 | 0 | 0 | 1 | 0 | 0
  HgL, Within, Below: number analyzed (Participants) | 7 | 8 | 15 | 10 | 10 | 16
  HgL, Within, Below | 1 | 1 | 0 | 0 | 1 | 2
  HgL, Within, Within: number analyzed (Participants) | 7 | 8 | 15 | 10 | 10 | 16
  HgL, Within, Within | 6 | 7 | 14 | 9 | 8 | 14
  HgL, Within, Above: number analyzed (Participants) | 7 | 8 | 15 | 10 | 10 | 16
  HgL, Within, Above | 0 | 0 | 1 | 0 | 1 | 0
  HgL, Above, Within: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 1
  HgL, Above, Within | 0 | 0 | 0 | 0 | 0 | 1
  HgL, Above, Above: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 1
  HgL, Above, Above | 0 | 0 | 1 | 0 | 0 | 0
  WBC, Below, Within: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 1
  WBC, Below, Within | 0 | 0 | 1 | 0 | 0 | 1
  WBC, Within, Unknown: number analyzed (Participants) | 10 | 10 | 14 | 11 | 7 | 16
  WBC, Within, Unknown | 0 | 0 | 0 | 1 | 0 | 0
  WBC, Within, Below: number analyzed (Participants) | 10 | 10 | 14 | 11 | 7 | 16
  WBC, Within, Below | 1 | 2 | 3 | 0 | 1 | 2
  WBC, Within, Within: number analyzed (Participants) | 10 | 10 | 14 | 11 | 7 | 16
  WBC, Within, Within | 9 | 7 | 11 | 10 | 5 | 14
  WBC, Within, Above: number analyzed (Participants) | 10 | 10 | 14 | 11 | 7 | 16
  WBC, Within, Above | 0 | 1 | 0 | 0 | 1 | 0
  WBC, Above, Within: number analyzed (Participants) | 0 | 0 | 2 | 0 | 3 | 0
  WBC, Above, Within | 0 | 0 | 1 | 0 | 2 | 0
  WBC, Above, Above: number analyzed (Participants) | 0 | 0 | 2 | 0 | 3 | 0
  WBC, Above, Above | 0 | 0 | 1 | 0 | 1 | 0
  PLC, Within, Unknown: number analyzed (Participants) | 10 | 9 | 15 | 9 | 5 | 15
  PLC, Within, Unknown | 0 | 0 | 0 | 1 | 0 | 0
  PLC, Within, Below: number analyzed (Participants) | 10 | 9 | 15 | 9 | 5 | 15
  PLC, Within, Below | 0 | 1 | 0 | 0 | 0 | 0
  PLC, Within, Within: number analyzed (Participants) | 10 | 9 | 15 | 9 | 5 | 15
  PLC, Within, Within | 10 | 7 | 15 | 7 | 4 | 14
  PLC, Within, Above: number analyzed (Participants) | 10 | 9 | 15 | 9 | 5 | 15
  PLC, Within, Above | 0 | 1 | 0 | 1 | 1 | 1
  PLC, Above, Within: number analyzed (Participants) | 0 | 1 | 2 | 2 | 5 | 2
  PLC, Above, Within | 0 | 1 | 2 | 2 | 4 | 1
  PLC, Above, Above: number analyzed (Participants) | 0 | 1 | 2 | 2 | 5 | 2
  PLC, Above, Above | 0 | 0 | 0 | 0 | 1 | 1

10. Primary Outcome: Number of Subjects With Hematological Laboratory Results Change With Respect to Normal Laboratory Ranges and Versus Baseline, at Day 38
Description: Assessed hematological laboratory parameters include hemoglobin level [HgL] white blood cells [WBC] and platelet count [PLC]. Hematological abnormalities refer to range indicator at timing, categorized as Below, Within or Above normal ranges, and compared to baseline range indicator of the same parameter, at Screening (Day-29 to Day 1) i.e. Below, Within or Above. [e.g. HgL, Below, Below = HgL below normal ranges at baseline versus below normal ranges at Day 38].
Time Frame: At Day 38
Population: This analysis was performed on the Exposed Set, which included all subjects with at least one study vaccine administration documented and with available results for the specified parameter and time point.
  As per Protocol, hematology testing for RSV HD group on Day 38 was not performed since no platelet decrease (i.e. less than 150000 cells/cubic millimeter) was detected on Day 32.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV LD Group | RSV MD Group | RSV HD Group | Placebo LD Group | Placebo MD Group | Placebo HD Group
Number analyzed (Participants) | 8 | 1 | 0 | 6 | 2 | 2
Participants
  HgL, Below, Below: number analyzed (Participants) | 2 | 0 | 0 | 1 | 0 | 0
  HgL, Below, Below | 2 | 0 | 0 | 1 | 0 | 0
  HgL, Within, Within: number analyzed (Participants) | 6 | 1 | 0 | 5 | 2 | 1
  HgL, Within, Within | 6 | 1 | 0 | 5 | 2 | 1
  HgL, Above, Above: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  HgL, Above, Above | 0 | 0 | 0 | 0 | 0 | 1
  WBC, Within, Within: number analyzed (Participants) | 8 | 1 | 0 | 6 | 1 | 2
  WBC, Within, Within | 8 | 1 | 0 | 4 | 1 | 2
  WBC, Within, Above: number analyzed (Participants) | 8 | 1 | 0 | 6 | 1 | 2
  WBC, Within, Above | 0 | 0 | 0 | 2 | 0 | 0
  WBC, Above, Above: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  WBC, Above, Above | 0 | 0 | 0 | 0 | 1 | 0
  PLC, Within, Within: number analyzed (Participants) | 8 | 1 | 0 | 6 | 1 | 2
  PLC, Within, Within | 7 | 1 | 0 | 5 | 0 | 1
  PLC, Within, Above: number analyzed (Participants) | 8 | 1 | 0 | 6 | 1 | 2
  PLC, Within, Above | 1 | 0 | 0 | 1 | 1 | 1
  PLC, Above, Above: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  PLC, Above, Above | 0 | 0 | 0 | 0 | 1 | 0

11. Primary Outcome: Number of Subjects With Hematological Laboratory Results Change With Respect to Normal Laboratory Ranges and Versus Baseline, at Day 61
Description: Assessed hematological laboratory parameters include hemoglobin level [HgL] white blood cells [WBC] and platelet count [PLC]. Hematological abnormalities refer to range indicator at timing, categorized as Below, Within or Above normal ranges, and compared to baseline range indicator of the same parameter, at Screening (Day-29 to Day 1) i.e. Unknown, Below, Within or Above. [e.g. HgL, Below, Below = HgL below normal ranges at baseline versus below normal ranges at Day 61].
Time Frame: At Day 61
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | RSV LD Group | RSV MD Group | RSV HD Group | Placebo LD Group | Placebo MD Group | Placebo HD Group
Number analyzed (Participants) | 10 | 12 | 16 | 9 | 11 | 15
Participants
  HgL, Below, Below: number analyzed (Participants) | 3 | 1 | 1 | 0 | 0 | 0
  HgL, Below, Below | 2 | 1 | 0 | 0 | 0 | 0
  HgL, Below, Within: number analyzed (Participants) | 3 | 1 | 1 | 0 | 0 | 0
  HgL, Below, Within | 1 | 0 | 1 | 0 | 0 | 0
  HgL, Within, Unknown: number analyzed (Participants) | 7 | 11 | 16 | 9 | 11 | 15
  HgL, Within, Unknown | 0 | 0 | 0 | 1 | 0 | 0
  HgL, Within, Below: number analyzed (Participants) | 7 | 11 | 16 | 9 | 11 | 15
  HgL, Within, Below | 0 | 1 | 0 | 0 | 0 | 2
  HgL, Within, Within: number analyzed (Participants) | 7 | 11 | 16 | 9 | 11 | 15
  HgL, Within, Within | 7 | 10 | 16 | 8 | 11 | 13
  HgL, Above, Within: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 1
  HgL, Above, Within | 0 | 0 | 0 | 0 | 0 | 1
  HgL, Above, Above: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 1
  HgL, Above, Above | 0 | 0 | 1 | 0 | 0 | 0
  WBC, Below, Within: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 1
  WBC, Below, Within | 0 | 0 | 1 | 0 | 0 | 1
  WBC, Within, Unknown: number analyzed (Participants) | 10 | 12 | 15 | 9 | 7 | 15
  WBC, Within, Unknown | 0 | 0 | 0 | 1 | 0 | 0
  WBC, Within, Below: number analyzed (Participants) | 10 | 12 | 15 | 9 | 7 | 15
  WBC, Within, Below | 1 | 0 | 0 | 0 | 0 | 3
  WBC, Within, Within: number analyzed (Participants) | 10 | 12 | 15 | 9 | 7 | 15
  WBC, Within, Within | 9 | 11 | 14 | 8 | 6 | 10
  WBC, Within, Above: number analyzed (Participants) | 10 | 12 | 15 | 9 | 7 | 15
  WBC, Within, Above | 0 | 1 | 1 | 0 | 1 | 2
  WBC, Above, Within: number analyzed (Participants) | 0 | 0 | 2 | 0 | 4 | 0
  WBC, Above, Within | 0 | 0 | 1 | 0 | 4 | 0
  WBC, Above, Above: number analyzed (Participants) | 0 | 0 | 2 | 0 | 4 | 0
  WBC, Above, Above | 0 | 0 | 1 | 0 | 0 | 0
  PLC, Within, Unknown: number analyzed (Participants) | 10 | 11 | 16 | 6 | 6 | 14
  PLC, Within, Unknown | 0 | 0 | 0 | 1 | 0 | 0
  PLC, Within, Below: number analyzed (Participants) | 10 | 11 | 16 | 6 | 6 | 14
  PLC, Within, Below | 0 | 0 | 0 | 0 | 0 | 1
  PLC, Within, Within: number analyzed (Participants) | 10 | 11 | 16 | 6 | 6 | 14
  PLC, Within, Within | 9 | 8 | 15 | 4 | 5 | 8
  PLC, Within, Above: number analyzed (Participants) | 10 | 11 | 16 | 6 | 6 | 14
  PLC, Within, Above | 1 | 3 | 1 | 1 | 1 | 5
  PLC, Above, Within: number analyzed (Participants) | 0 | 1 | 2 | 2 | 5 | 2
  PLC, Above, Within | 0 | 1 | 2 | 2 | 4 | 1
  PLC, Above, Above: number analyzed (Participants) | 0 | 1 | 2 | 2 | 5 | 2
  PLC, Above, Above | 0 | 0 | 0 | 0 | 1 | 1

12. Primary Outcome: Number of Subjects With Biochemical Laboratory Results Change With Respect to Normal Laboratory Ranges and Versus Baseline, at Day 31
Description: Assessed biochemical laboratory parameters include alanine aminotransferase [ALT], aspartate aminotransferase [AST] and creatinine [CREA]. Biochemical abnormalities refer to range indicator at timing, categorized as Below, Within or Above normal ranges, and compared to baseline range indicator of the same parameter, at Screening (Day-29 to Day 1) i.e. Unknown, Below, Within or Above. [e.g. ALT, Below, Below = ALT below normal ranges at baseline versus below normal ranges at Day 31].
Time Frame: At Day 31
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | RSV LD Group | RSV MD Group | RSV HD Group | Placebo LD Group | Placebo MD Group | Placebo HD Group
Number analyzed (Participants) | 9 | 11 | 16 | 11 | 9 | 17
Participants
  ALT, Below, Below: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 1
  ALT, Below, Below | 1 | 0 | 0 | 0 | 0 | 0
  ALT, Below, Within: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 1
  ALT, Below, Within | 1 | 0 | 0 | 0 | 0 | 0
  ALT, Below, Above: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 1
  ALT, Below, Above | 0 | 0 | 0 | 0 | 0 | 1
  ALT, Within, Unknown: number analyzed (Participants) | 8 | 11 | 16 | 11 | 9 | 13
  ALT, Within, Unknown | 0 | 1 | 0 | 0 | 0 | 0
  ALT, Within, Below: number analyzed (Participants) | 8 | 11 | 16 | 11 | 9 | 13
  ALT, Within, Below | 1 | 0 | 0 | 0 | 0 | 0
  ALT, Within, Within: number analyzed (Participants) | 8 | 11 | 16 | 11 | 9 | 13
  ALT, Within, Within | 7 | 10 | 15 | 11 | 7 | 13
  ALT, Within, Above: number analyzed (Participants) | 8 | 11 | 16 | 11 | 9 | 13
  ALT, Within, Above | 0 | 0 | 1 | 0 | 2 | 0
  ALT, Above, Within: number analyzed (Participants) | 0 | 1 | 2 | 0 | 0 | 3
  ALT, Above, Within | 0 | 1 | 1 | 0 | 0 | 2
  ALT, Above, Above: number analyzed (Participants) | 0 | 1 | 2 | 0 | 0 | 3
  ALT, Above, Above | 0 | 0 | 1 | 0 | 0 | 1
  AST, Within, Unknown: number analyzed (Participants) | 9 | 9 | 15 | 10 | 8 | 14
  AST, Within, Unknown | 0 | 1 | 0 | 0 | 0 | 0
  AST, Within, Within: number analyzed (Participants) | 9 | 9 | 15 | 10 | 8 | 14
  AST, Within, Within | 9 | 7 | 13 | 9 | 7 | 14
  AST, Within, Above: number analyzed (Participants) | 9 | 9 | 15 | 10 | 8 | 14
  AST, Within, Above | 0 | 1 | 2 | 1 | 1 | 0
  AST, Above, Below: number analyzed (Participants) | 1 | 3 | 3 | 1 | 1 | 3
  AST, Above, Below | 0 | 0 | 0 | 0 | 0 | 1
  AST, Above, Within: number analyzed (Participants) | 1 | 3 | 3 | 1 | 1 | 3
  AST, Above, Within | 1 | 1 | 1 | 1 | 0 | 0
  AST, Above, Above: number analyzed (Participants) | 1 | 3 | 3 | 1 | 1 | 3
  AST, Above, Above | 0 | 2 | 2 | 0 | 1 | 2
  CREA, Below, Unknown: number analyzed (Participants) | 7 | 4 | 4 | 8 | 1 | 0
  CREA, Below, Unknown | 0 | 1 | 0 | 0 | 0 | 0
  CREA, Below, Below: number analyzed (Participants) | 7 | 4 | 4 | 8 | 1 | 0
  CREA, Below, Below | 4 | 3 | 1 | 7 | 1 | 0
  CREA, Below, Within: number analyzed (Participants) | 7 | 4 | 4 | 8 | 1 | 0
  CREA, Below, Within | 3 | 0 | 3 | 1 | 0 | 0
  CREA, Within, Below: number analyzed (Participants) | 3 | 8 | 14 | 3 | 7 | 17
  CREA, Within, Below | 3 | 1 | 4 | 0 | 0 | 4
  CREA, Within, Within: number analyzed (Participants) | 3 | 8 | 14 | 3 | 7 | 17
  CREA, Within, Within | 0 | 7 | 10 | 3 | 7 | 12
  CREA, Within, Above: number analyzed (Participants) | 3 | 8 | 14 | 3 | 7 | 17
  CREA, Within, Above | 0 | 0 | 0 | 0 | 0 | 1
  CREA, Above, Within: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  CREA, Above, Within | 0 | 0 | 0 | 0 | 1 | 0

13. Primary Outcome: Number of Subjects With Biochemical Laboratory Results Change With Respect to Normal Laboratory Ranges and Versus Baseline, at Day 61
Description: Assessed biochemical laboratory parameters include alanine aminotransferase [ALT], aspartate aminotransferase [AST] and creatinine [CREA]. Biochemical abnormalities refer to range indicator at timing, categorized as Below, Within or Above normal ranges, and compared to baseline range indicator of the same parameter, at Screening (Day-29 to Day 1) i.e. Below, Within or Above. [e.g. ALT, Below, Below = ALT below normal ranges at baseline versus below normal ranges at Day 61].
Time Frame: At Day 61
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | RSV LD Group | RSV MD Group | RSV HD Group | Placebo LD Group | Placebo MD Group | Placebo HD Group
Number analyzed (Participants) | 9 | 11 | 16 | 11 | 10 | 16
Participants
  ALT, Below, Below: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 1
  ALT, Below, Below | 1 | 0 | 0 | 0 | 0 | 0
  ALT, Below, Within: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 1
  ALT, Below, Within | 1 | 0 | 0 | 0 | 0 | 1
  ALT, Within, Within: number analyzed (Participants) | 8 | 11 | 16 | 11 | 10 | 12
  ALT, Within, Within | 8 | 10 | 15 | 10 | 9 | 12
  ALT, Within, Above: number analyzed (Participants) | 8 | 11 | 16 | 11 | 10 | 12
  ALT, Within, Above | 0 | 1 | 1 | 1 | 1 | 0
  ALT, Above, Within: number analyzed (Participants) | 0 | 1 | 2 | 0 | 1 | 2
  ALT, Above, Within | 0 | 1 | 2 | 0 | 1 | 1
  ALT, Above, Above: number analyzed (Participants) | 0 | 1 | 2 | 0 | 1 | 2
  ALT, Above, Above | 0 | 0 | 0 | 0 | 0 | 1
  AST, Within, Within: number analyzed (Participants) | 9 | 10 | 15 | 10 | 9 | 13
  AST, Within, Within | 9 | 9 | 15 | 10 | 8 | 13
  AST, Within, Above: number analyzed (Participants) | 9 | 10 | 15 | 10 | 9 | 13
  AST, Within, Above | 0 | 1 | 0 | 0 | 1 | 0
  AST, Above, Within: number analyzed (Participants) | 1 | 2 | 3 | 1 | 2 | 3
  AST, Above, Within | 1 | 1 | 1 | 0 | 0 | 1
  AST, Above, Above: number analyzed (Participants) | 1 | 2 | 3 | 1 | 2 | 3
  AST, Above, Above | 0 | 1 | 2 | 1 | 2 | 2
  CREA, Below, Below: number analyzed (Participants) | 7 | 3 | 4 | 8 | 2 | 0
  CREA, Below, Below | 4 | 2 | 2 | 7 | 1 | 0
  CREA, Below, Within: number analyzed (Participants) | 7 | 3 | 4 | 8 | 2 | 0
  CREA, Below, Within | 3 | 1 | 2 | 1 | 1 | 0
  CREA, Within, Below: number analyzed (Participants) | 3 | 9 | 14 | 3 | 8 | 16
  CREA, Within, Below | 3 | 1 | 3 | 0 | 0 | 1
  CREA, Within, Within: number analyzed (Participants) | 3 | 9 | 14 | 3 | 8 | 16
  CREA, Within, Within | 0 | 8 | 10 | 3 | 8 | 15
  CREA, Within, Above: number analyzed (Participants) | 3 | 9 | 14 | 3 | 8 | 16
  CREA, Within, Above | 0 | 0 | 1 | 0 | 0 | 0
  CREA, Above, Within: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  CREA, Above, Within | 0 | 0 | 0 | 0 | 1 | 0

14. Secondary Outcome: Number of Subjects With Any SAEs From Day 1 up to Day 366
Description: as for outcome 4
Time Frame: From Day 1 up to Day 366
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | RSV LD Group | RSV MD Group | RSV HD Group | Placebo LD Group | Placebo MD Group | Placebo HD Group
Number analyzed (Participants) | 11 | 14 | 18 | 11 | 11 | 17
Participants | 1 | 1 | 1 | 3 | 1 | 2

15. Secondary Outcome: Number of Subjects With Lower Respiratory Tract Infection Associated With RSV Infection (RSV-LRTI) (AE of Specific Interest) From Dose 1 Administration (Day 1) up to Day 366
Description: Subjects experiencing an LRTI associated with RSV infection were reported as AE of specific interest. To identify RSV-LRTI for the purpose of AE of specific interest, the diagnosis was based on the investigators' clinical judgment taking into account the clinical history, the examination, relevant medical investigations and locally-available diagnostic test for RSV.
Time Frame: From Dose 1 administration (Day 1) up to Day 366
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | RSV LD Group | RSV MD Group | RSV HD Group | Placebo LD Group | Placebo MD Group | Placebo HD Group
Number analyzed (Participants) | 11 | 14 | 18 | 11 | 11 | 17
Participants | 0 | 1 | 0 | 3 | 0 | 0

16. Secondary Outcome: Number of Subjects With Respiratory Tract Infection Associated With RSV Infection (RSV-RTI), RSV-LRTI, Severe RSV-LRTI (According to Standardized Case Definitions) From Dose 1 Administration (Day 1) up to Day 366
Description: RSV-RTI refers to subject having runny nose OR blocked nose OR cough AND confirmed RSV infection [RSV infection confirmed on nasal swab positive for RSV A or B by quantitative Reverse Transcription Polymerase Chain Reaction (qRT-PCR) performed at sponsor level]. RSV-LRTI refers to subject with history of cough OR difficulty breathing [based on history reported by parents/legally acceptable representatives (LARs) and includes difficulty breathing (e.g. showing signs of wheezing or stridor, tachypnoea, flaring of nostrils, chest in-drawing, apnoea) associated with nasal obstruction] AND Blood Oxygen Saturation (SpO2) lower than (<) 95 percent (%), OR respiratory rate (RR) increase [defined as ≥ 40/minute (12 months of age or above)] AND confirmed RSV infection. RSV-severe LRTI are cases meeting the case definition of RSV-LRTI AND SpO2 < 93%, OR lower chest wall in-drawing.
Time Frame: From Dose 1 administration (Day 1) up to Day 366
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | RSV LD Group | RSV MD Group | RSV HD Group | Placebo LD Group | Placebo MD Group | Placebo HD Group
Number analyzed (Participants) | 11 | 14 | 18 | 11 | 11 | 17
Participants
  RSV-RTI | 1 | 3 | 1 | 4 | 3 | 3
  RSV-LRTI | 0 | 0 | 0 | 1 | 0 | 0
  RSV-severe LRTI | 0 | 0 | 0 | 1 | 0 | 0

17. Secondary Outcome: Number of Subjects With Any SAEs From Day 1 up to Study Conclusion at Day 731
Description: as for outcome 4
Time Frame: From Day 1 up to study conclusion at Day 731
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | RSV LD Group | RSV MD Group | RSV HD Group | Placebo LD Group | Placebo MD Group | Placebo HD Group
Number analyzed (Participants) | 11 | 14 | 18 | 11 | 11 | 17
Participants | 1 | 1 | 2 | 3 | 1 | 2

18. Secondary Outcome: Number of Subjects With RSV-LRTI (AE of Specific Interest) From Dose 1 Administration (Day 1) up to Study Conclusion at Day 731
Description: as for outcome 15
Time Frame: From Dose 1 administration (Day 1) up to study conclusion at Day 731
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | RSV LD Group | RSV MD Group | RSV HD Group | Placebo LD Group | Placebo MD Group | Placebo HD Group
Number analyzed (Participants) | 11 | 14 | 18 | 11 | 11 | 17
Participants | 0 | 1 | 0 | 3 | 0 | 0

19. Secondary Outcome: Number of Subjects With RSV-RTI, RSV-LRTI, Severe RSV-LRTI (According to Standardized Case Definitions) From Dose 1 Administration (Day 1) up to Study Conclusion at Day 731
Description: RSV-RTI refers to subject having runny nose OR blocked nose OR cough AND confirmed RSV infection (RSV infection confirmed on nasal swab positive for RSV A or B by qRT-PCR performed at sponsor level). RSV-LRTI refers to subject with history of cough OR difficulty breathing [based on history reported by parents/LARs and includes difficulty breathing (e.g. showing signs of wheezing or stridor, tachypnoea, flaring of nostrils, chest in-drawing, apnoea) associated with nasal obstruction] AND Sp02 < 95% OR respiratory rate (RR) increase [defined as ≥ 40/minute (12 months of age or above)] AND confirmed RSV infection. RSV-severe LRTI are cases meeting the case definition of RSV-LRTI AND SpO2 < 93%, OR lower chest wall in-drawing.
Time Frame: From Dose 1 administration (Day 1) up to study conclusion at Day 731
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | RSV LD Group | RSV MD Group | RSV HD Group | Placebo LD Group | Placebo MD Group | Placebo HD Group
Number analyzed (Participants) | 11 | 14 | 18 | 11 | 11 | 17
Participants
  RSV-RTI | 2 | 6 | 2 | 5 | 4 | 4
  RSV-LRTI | 0 | 0 | 0 | 1 | 0 | 0
  RSV-severe LRTI | 0 | 0 | 0 | 1 | 0 | 0

20. Secondary Outcome: Frequency of RSV-specific CD4+ T-cells Expressing at Least Two Markers Upon Stimulation With F, N and M2-1 Peptide Pools
Description: Magnitude of cell mediated immunity (CMI) response to the investigational RSV vaccine was measured in terms of frequency of RSV-specific CD4+ T-cells expressing at least two markers upon stimulation with F, N and M2-1 peptide pools and expressed in RSV-specific CD4+ T-cells/million cells.
  Assessed markers were CD40-L, IL-2, TNF-α and IFN-ɣ.
Time Frame: At Pre-vaccination (Screening), Day 31, Day 61 and Day 366
Population: This analysis was performed on the Per-protocol set (PPS), which included all vaccinated subjects, meeting all protocol requirements and with available CMI results at the specified time point.
Measure: Median (Inter-Quartile Range); unit: RSV-specific CD4+ T-cells/million cells
Arm/Group | RSV LD Group | RSV MD Group | RSV HD Group | Placebo LD Group | Placebo MD Group | Placebo HD Group
Number analyzed (Participants) | 9 | 3 | 1 | 10 | 2 | 1
RSV-specific CD4+ T-cells/million cells
  RSV F pool 15/11 Ag, Screening: number analyzed (Participants) | 8 | 3 | 1 | 9 | 1 | 0
  RSV F pool 15/11 Ag, Screening | 169.5 [85 to 218] | 123 [32 to 268] | 1 [1 to 1] | 176 [120 to 336] | 1813 [1813 to 1813] |
  RSV F pool 15/11 Ag, Day 31: number analyzed (Participants) | 9 | 2 | 1 | 7 | 2 | 0
  RSV F pool 15/11 Ag, Day 31 | 291 [231 to 469] | 546 [484 to 608] | 1086 [1086 to 1086] | 234 [48 to 350] | 1129.5 [379 to 1880] |
  RSV F pool 15/11 Ag, Day 61: number analyzed (Participants) | 8 | 3 | 1 | 10 | 2 | 0
  RSV F pool 15/11 Ag, Day 61 | 214 [74.5 to 331.5] | 451 [93 to 495] | 394 [394 to 394] | 105.5 [1 to 193] | 759 [218 to 1300] |
  RSV F pool 15/11 Ag, Day 366: number analyzed (Participants) | 4 | 2 | 1 | 4 | 2 | 1
  RSV F pool 15/11 Ag, Day 366 | 206 [71 to 288.5] | 108.5 [1 to 216] | 1164 [1164 to 1164] | 252.5 [169.5 to 495] | 664.5 [252 to 1077] | 229 [229 to 229]
  RSV N pool 15/11 Ag, Screening: number analyzed (Participants) | 8 | 3 | 1 | 8 | 1 | 0
  RSV N pool 15/11 Ag, Screening | 51 [1 to 121] | 54 [1 to 369] | 140 [140 to 140] | 104 [27 to 174] | 253 [253 to 253] |
  RSV N pool 15/11 Ag, Day 31: number analyzed (Participants) | 8 | 2 | 1 | 9 | 2 | 0
  RSV N pool 15/11 Ag, Day 31 | 129.5 [23.5 to 226.5] | 229 [1 to 457] | 289 [289 to 289] | 58 [1 to 102] | 193 [180 to 206] |
  RSV N pool 15/11 Ag, Day 61: number analyzed (Participants) | 7 | 3 | 1 | 10 | 2 | 0
  RSV N pool 15/11 Ag, Day 61 | 70 [1 to 165] | 144 [34 to 426] | 1 [1 to 1] | 71 [50 to 117] | 64.5 [52 to 77] |
  RSV N pool 15/11 Ag, Day 366: number analyzed (Participants) | 6 | 2 | 1 | 6 | 2 | 1
  RSV N pool 15/11 Ag, Day 366 | 56 [1 to 269] | 41.5 [1 to 82] | 82 [82 to 82] | 89 [42 to 113] | 78 [27 to 129] | 91 [91 to 91]
  RSV M2-1 pool 15/11 Ag, Screening: number analyzed (Participants) | 5 | 3 | 1 | 5 | 1 | 0
  RSV M2-1 pool 15/11 Ag, Screening | 1 [1 to 9] | 1 [1 to 10] | 56 [56 to 56] | 1 [1 to 1] | 214 [214 to 214] |
  RSV M2-1 pool 15/11 Ag, Day 31: number analyzed (Participants) | 5 | 2 | 1 | 8 | 2 | 0
  RSV M2-1 pool 15/11 Ag, Day 31 | 1 [1 to 34] | 21.5 [1 to 42] | 229 [229 to 229] | 1 [1 to 13] | 145.5 [100 to 191] |
  RSV M2-1 pool 15/11 Ag, Day 61: number analyzed (Participants) | 6 | 3 | 1 | 9 | 2 | 0
  RSV M2-1 pool 15/11 Ag, Day 61 | 8 [1 to 57] | 2 [1 to 55] | 46 [46 to 46] | 30 [1 to 33] | 1 [1 to 1] |
  RSV M2-1 pool 15/11 Ag, Day 366: number analyzed (Participants) | 6 | 2 | 1 | 5 | 2 | 1
  RSV M2-1 pool 15/11 Ag, Day 366 | 7 [1 to 81] | 2.5 [1 to 4] | 13 [13 to 13] | 23 [6 to 27] | 48 [1 to 95] | 56 [56 to 56]

21. Secondary Outcome: Anti-RSV-A Neutralizing Antibody Titers
Description: Humoral response to the investigational RSV vaccine was measured in terms of anti-RSV-A neutralizing antibody titers and expressed as geometric mean titers (GMTs) in Estimated Dilution 60 (ED60) titers.
Time Frame: At Pre-vaccination (Screening), Day 31, Day 61 and Day 366
Population: This analysis was performed on the Per-protocol set (PPS), which included all vaccinated subjects, meeting all protocol requirements and with available immunogenicity results for the specified assay and time point.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | RSV LD Group | RSV MD Group | RSV HD Group | Placebo LD Group | Placebo MD Group | Placebo HD Group
Number analyzed (Participants) | 10 | 13 | 18 | 11 | 11 | 17
Titers
  Screening: number analyzed (Participants) | 10 | 13 | 17 | 10 | 11 | 16
  Screening | 127.4 [44 to 368.5] | 179.4 [99.2 to 324.5] | 495.7 [242.5 to 1013.1] | 376.5 [89.3 to 1587.5] | 214.6 [80.8 to 569.9] | 332 [158.5 to 695.4]
  Day 31: number analyzed (Participants) | 10 | 12 | 18 | 10 | 9 | 17
  Day 31 | 711.7 [229.7 to 2204.9] | 1646 [815.8 to 3321] | 2203.9 [1383.7 to 3510.3] | 645.9 [266.3 to 1566.5] | 703.9 [244.3 to 2028.4] | 295 [149.6 to 581.8]
  Day 61: number analyzed (Participants) | 10 | 12 | 17 | 11 | 11 | 15
  Day 61 | 1081.3 [648.3 to 1803.3] | 1809 [1022.6 to 3200.2] | 1974.9 [1356.9 to 2874.3] | 421.5 [178.9 to 993.1] | 316.4 [169 to 592.3] | 307.1 [148.5 to 634.9]
  Day 366: number analyzed (Participants) | 9 | 11 | 16 | 11 | 11 | 16
  Day 366 | 236.9 [105.7 to 531] | 837 [546.6 to 1281.6] | 1038 [629.3 to 1712.3] | 398.5 [163.5 to 971.7] | 545.4 [269.4 to 1104.3] | 493.8 [216 to 1129.1]

22. Secondary Outcome: Anti-RSV-F Antibody Concentrations
Description: Humoral response to the investigational RSV vaccine was measured as anti-RSV F antibody concentrations and expressed as geometric mean concentrations (GMCs) in enzyme-linked immunosorbent assay (ELISA) units per milliliter (EU/mL).
Time Frame: At Pre-vaccination (Screening), Day 31, Day 61 and Day 366
Population: as for outcome 21
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | RSV LD Group | RSV MD Group | RSV HD Group | Placebo LD Group | Placebo MD Group | Placebo HD Group
Number analyzed (Participants) | 10 | 13 | 17 | 11 | 11 | 17
EU/mL
  Screening: number analyzed (Participants) | 9 | 13 | 17 | 10 | 9 | 16
  Screening | 2082 [864.3 to 5015.5] | 2061.6 [1343.6 to 3163.4] | 3686.4 [1964.5 to 6917.5] | 3933.2 [1789.1 to 8646.7] | 1216.3 [472.9 to 3128.7] | 2988.6 [1420.9 to 6286]
  Day 31: number analyzed (Participants) | 10 | 11 | 17 | 9 | 9 | 17
  Day 31 | 4807.2 [1738.5 to 13292.8] | 10810.9 [4062.2 to 28771.1] | 17419 [11639.6 to 26068.2] | 6134.2 [2752 to 13673] | 7911.6 [3187.7 to 19636] | 2350.6 [1235.9 to 4470.7]
  Day 61: number analyzed (Participants) | 9 | 12 | 15 | 11 | 11 | 15
  Day 61 | 6167.5 [3701.3 to 10277.1] | 15577.4 [8012.9 to 30283.2] | 15083.8 [10555 to 21555.7] | 2983.3 [1612.8 to 5518.3] | 3182 [1737.1 to 5828.8] | 2101.3 [1038.3 to 4252.6]
  Day 366: number analyzed (Participants) | 9 | 11 | 17 | 11 | 11 | 16
  Day 366 | 3988.5 [1789.4 to 8890.1] | 6521.1 [3702.5 to 11485.4] | 6490.7 [4509.7 to 9341.8] | 3591.3 [1472.8 to 8756.9] | 3047.5 [1577.7 to 5886.6] | 4487.9 [1936.8 to 10398.8]

23. Secondary Outcome: Palivizumab-competing Antibody Concentrations
Description: Humoral response to the investigational RSV vaccine was measured as Palivizumab-competing antibody concentrations and expressed as geometric mean concentrations (GMCs) in microgram/milliliter (µg/mL).
Time Frame: At Pre-vaccination (Screening), Day 31 and Day 61
Population: as for outcome 21
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | RSV LD Group | RSV MD Group | RSV HD Group | Placebo LD Group | Placebo MD Group | Placebo HD Group
Number analyzed (Participants) | 10 | 13 | 17 | 11 | 11 | 17
µg/mL
  Screening: number analyzed (Participants) | 9 | 13 | 17 | 10 | 9 | 16
  Screening | 5.2 [4.3 to 6.3] | 4.8 [4.8 to 4.8] | 6.6 [5 to 8.6] | 6.2 [4.2 to 9.2] | 4.8 [4.8 to 4.8] | 7.2 [4.8 to 10.9]
  Day 31: number analyzed (Participants) | 10 | 11 | 17 | 9 | 9 | 17
  Day 31 | 7.9 [5.3 to 11.7] | 11.1 [6.2 to 19.8] | 17.5 [13 to 23.6] | 8 [4.4 to 14.5] | 12.5 [6.2 to 25.5] | 6.8 [4.8 to 9.6]
  Day 61: number analyzed (Participants) | 9 | 12 | 15 | 11 | 11 | 15
  Day 61 | 6.3 [4.6 to 8.6] | 15.2 [9.2 to 25.1] | 14 [10.1 to 19.4] | 6.1 [4.3 to 8.6] | 7 [4.5 to 10.8] | 6.6 [4.8 to 9]

ADVERSE EVENTS:
Time Frame: Solicited adverse events were collected during the 7-day follow-up period and unsolicited adverse events during the 30-day follow-up period after any vaccination. Serious adverse events were collected from Day 1 up to Day 731.
Arm/Group | RSV LD Group | RSV MD Group | RSV HD Group | Placebo LD Group | Placebo MD Group | Placebo HD Group
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/14 | 0/18 | 0/11 | 0/11 | 0/17
Serious Adverse Events (participants affected / at risk) | 1/11 | 1/14 | 2/18 | 3/11 | 1/11 | 2/17
Other Adverse Events (participants affected / at risk) | 10/11 | 11/14 | 17/18 | 11/11 | 10/11 | 14/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RSV LD Group (N=11) | RSV MD Group (N=14) | RSV HD Group (N=18) | Placebo LD Group (N=11) | Placebo MD Group (N=11) | Placebo HD Group (N=17)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Coronavirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpangina (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Unresponsive to stimuli (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RSV LD Group (N=11) | RSV MD Group (N=14) | RSV HD Group (N=18) | Placebo LD Group (N=11) | Placebo MD Group (N=11) | Placebo HD Group (N=17)
Pyrexia (General disorders) | 5 (7) | 5 (5) | 11 (15) | 5 (5) | 4 (6) | 2 (2)
Injection site erythema (General disorders) | 2 (4) | 2 (2) | 4 (5) | 3 (6) | 0 (0) | 4 (5)
Injection site pain (General disorders) | 3 (3) | 3 (4) | 2 (2) | 2 (3) | 0 (0) | 4 (5)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 3 (4)
Nasopharyngitis (Infections and infestations) | 2 (2) | 6 (10) | 7 (8) | 0 (0) | 4 (5) | 5 (7)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 3 (3) | 1 (1)
Conjunctivitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Croup infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acarodermatitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (3) | 0 (0) | 2 (3) | 2 (3) | 3 (3)
Teething (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-12-10): https://cdn.clinicaltrials.gov/large-docs/73/NCT02927873/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-28): https://cdn.clinicaltrials.gov/large-docs/73/NCT02927873/SAP_001.pdf